CLINICAL TRIAL: NCT03669874
Title: Clinical Application of MUSE System for Ultrasound-guided Endoscopic Fundoplication for Gastro-esophageal Reflux Disease Patients
Brief Title: Endoscopic Fundoplication With MUSE System
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pier Alberto Testoni, Professor, IRCCS San Raffaele
Other Study IDs: MUSE/2015
Record Dates: First submitted 2018-08-30; First posted 2018-09-13 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Gastro-esophageal Reflux; Endoscopic Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Endoscopic fundoplication — Endoscopic fundoplication is a less invasive alternative to the traditional surgical fundoplication.
  The MUSE device is similar to an endoscope, so the whole procedure can be done by a single operator. The device is composed of a shaft with a distal rigid part which is placed in the esophagus 3 cm proximal to the esophago-gastric junction containing a cartridge holding five B-shaped titanium surgical Staples and a tip which is retroflexed and contains an ultrasonic transducer which defines the correct tissue thickness for stapling the fundus against the esophagus. The device must be extracted to be reloaded with 5 more staples at a time for creation of a 180° anterior fundoplication.

SUMMARY:
This is a spontaneous, prospective, monocentric, observational, cohort study, with the aim of evaluating the effect of ultrasound-guided endoscopic fundoplication using the Medigus Ultrasonic Surgical Endostapler (MUSESystem; MediGus, Ltd. Israel) in patients with esophageal or extra-esophageal gastro-oesophageal reflux disease (GERD)-related symptoms. The end of the study will be at the end of the 6-year follow-up of the last patient enrolled. The study proposes the following objectives:

* Primary objective: to evaluate the efficacy of endoscopic fundoplication with MUSE for the treatment of GERD, through clinical experience, in terms of:

  * effect on GERD-Health Related Quality of Life (HRQL) and Reflux Symptom Index (RSI) questionnaire scores
  * effect on the use and dosage of proton pump inhibitors (PPI)
  * feasibility and safety of the endoluminal fundoplication procedure
* Secondary objective: to characterize the treated patient population (demographic and objective data) and to identify the successful predictors of the procedure.

The study design includes the following phases:

*Preliminary patient evaluation and verification of inclusion criteria through: Upper GI endoscopy Esophageal high-resolution manometry 24-hours esophageal pH-impedance OFF PPI PPI use GERD-HRQL and RSI questionnaires scores OFF PPI

* 6-month follow-up: Upper GI endoscopy Esophageal high-resolution manometry 24-hours esophageal pH-impedance OFF PPI PPI use GERD-HRQL and RSI questionnaires scores OFF PPI
* 12-months follow-up: Upper GI endoscopy 24-hours esophageal pH-impedance OFF PPI PPI use GERD-HRQL and RSI questionnaires scores OFF PPI
* Yearly clinical follow-up (up to 6 years):

PPI use GERD-HRQL and RSI questionnaires scores OFF PPI

ELIGIBILITY:
Inclusion Criteria:

* Chronic (> 6 months) GERD-related esophageal or extra-esophageal symptoms
* Endoscopic or pH-impedance evidence of GERD (esophagitis, Barrett's esophagus, NERD, hypersensitive esophagus)
* Indication to surgical fundoplication
* Patients available for a long-term follow-up

Exclusion Criteria:

* Hiatal hernia ≥ 3 cm
* Major esophageal motility disorder
* Esophageal stenosis
* Malignant neoplasia (except minor superficial skin neoplasm)
* Portal hypertension, bleeding disorders so to controindicate surgery, esophageal varices, stenosis or diverticula
* Previous cardiac, thoracic or upper GI surgery
* BMI >40
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are selected from tertiary care center
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-09-16 (Actual); Primary Completion 2021-09-16 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 6 months
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 12 months
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 24 months
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 3 years
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 4 years
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 5 years
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in GERD-HRQL (Gastro-esophageal Reflux Disease-Health Related quality of life) questionnaire score | change from baseline GERD-HRQL at 6 years
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 6 months
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 12 months
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 24 months
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 3 years
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 4 years
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 5 years
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by change in RSI (Reflux Symptom Index) questionnaire score | change from baseline RSI at 6 years
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 6 months
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 12 months
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 24 months
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 3 years
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 4 years
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 5 years
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy
To evaluate clinical efficacy of endoscopic fundoplication with MUSE as assessed by changes in proton pump inhibitors (PPI) consumption | change from baseline PPI consumption at 6 years
  Gastric antisecretive therapy with proton pump inhibitors (PPI) is the gold standard for the treatment of GERD. This therapy is a chronic therapy with possible side effects. The endoscopic procedure under study aims to halved or discontinue the medical therapy

SECONDARY OUTCOMES:
To identify endoscopic factors predicting positive outcomes: changes in hiatal hernia size | change from baseline hiatal hernia size at 6 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The size of a hiatal hernia is a parameter describing the continence characteristics of the sphincter neo-valve.
To identify endoscopic factors predicting positive outcomes: changes in hiatal hernia size | change from baseline hiatal hernia size at 12 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The size of a hiatal hernia is a parameter describing the continence characteristics of the sphincter neo-valve.
To identify endoscopic factors predicting positive outcomes: changes in Hill's grade | change from baseline Hill's grade at 6 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The Hill's grade is a parameter describing the continence characteristics of the sphincter neo-valve. The Hill's grade range from I to IV; the higher grades represents worse outcomes (worse valve's continence).
To identify endoscopic factors predicting positive outcomes: changes in Hill's grade | change from baseline Hill's grade at 12 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The Hill's grade is a parameter describing the continence characteristics of the sphincter neo-valve. The Hill's grade range from I to IV; the higher grades represents worse outcomes (worse valve's continence).
To identify endoscopic factors predicting positive outcomes: changes in Jobe's lenght | change from baseline Jobe's lenght at 6 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The Jobe's lenght is a parameter describing the continence characteristics of the sphincter neo-valve.
To identify endoscopic factors predicting positive outcomes: changes in Jobe's lenght | change from baseline Jobe's lenght at 12 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The Jobe's lenght is a parameter describing the continence characteristics of the sphincter neo-valve.
To identify endoscopic factors predicting positive outcomes: changes in esophagitis' grade | change from baseline esophagitis' grade at 6 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The presence of esophagitis and its grade, as defined by the Los Angeles classification, is a parameter of procedure's efficacy. The esophagitis grade range from A to D; the higher grades represents worse outcomes.
To identify endoscopic factors predicting positive outcomes: changes in esophagitis' grade | change from baseline esophagitis' grade at 12 months
  Endoscopic fundoplication with MUSE modifies the anatomy of the esophago-gastric junction to reduce the reflux of gastric contents into the esophagus. The presence of esophagitis and its grade, as defined by the Los Angeles classification, is a parameter of procedure's efficacy. The esophagitis grade range from A to D; the higher grades represents worse outcomes.
To identify pathophysiological factors predicting positive outcomes: changes in DeMeester score | change from baseline DeMeester score at 6 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux. DeMeester score is a composite score which examined six variables (number of reflux episodes, number of episodes longer than 5 minutes, longest reflux duration, total percentage of monitoring time with pH below 4, and the percentage of time with pH below 4 in an upright position and supine position). A score of >14.72 shows a pathological reflux. Higher values represent worse outcomes.
To identify pathophysiological factors predicting positive outcomes: changes in DeMeester score | change from baseline DeMeester score at 12 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux. DeMeester score is a composite score which examined six variables (number of reflux episodes, number of episodes longer than 5 minutes, longest reflux duration, total percentage of monitoring time with pH below 4, and the percentage of time with pH below 4 in an upright position and supine position). A score of >14.72 shows a pathological reflux. Higher values represent worse outcomes.
To identify pathophysiological factors predicting positive outcomes: changes in AET (Acid Exposure Time) | change from baseline AET at 6 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in AET (Acid Exposure Time) | change from baseline AET at 12 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in longest reflux episode (min) | change from baseline longest reflux episode at 6 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in longest reflux episode (min) | change from baseline longest reflux episode at 12 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of refluxes greater than 5 minutes | change from baseline number of refluxes greater than 5 minutes at 6 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of refluxes greater than 5 minutes | change from baseline number of refluxes greater than 5 minutes at 12 months
  parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of total refluxes | change from baseline number of total refluxes at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of total refluxes | change from baseline number of total refluxes at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of acid refluxes | change from baseline number of acid refluxes at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of acid refluxes | change from baseline number of acid refluxes at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of weakly acid refluxes | change from baseline number of weakly acid refluxes at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of weakly acid refluxes | change from baseline number of weakly acid refluxes at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of not acid refluxes | change from baseline number of not acid refluxes at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of not acid refluxes | change from baseline number of not acid refluxes at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of proximal refluxes | change from baseline number of proximal refluxes at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in number of proximal refluxes | change from baseline number of proximal refluxes at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in MNBI (Mean Nocturnal Baseline Impedance) | change from baseline MNBI at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in MNBI (Mean Nocturnal Baseline Impedance) | change from baseline MNBI at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in PSPW (Post Swallow reflux-induced Peristaltic Waves) | change from baseline PSPW at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in PSPW (Post Swallow reflux-induced Peristaltic Waves) | change from baseline PSPW at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in BCT (Bolus Clearance Time) | change from baseline BCT at 6 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in BCT (Bolus Clearance Time) | change from baseline BCT at 12 months
  parameter detected by 24hours esophagel impedance. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
To identify pathophysiological factors predicting positive outcomes: changes in LES (Lower Esophageal Sphincter) basal pressure | change from baseline LES basal pressure at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in LES (Lower Esophageal Sphincter) basal pressure | change from baseline LES basal pressure at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in LES (Lower Esophageal Sphincter) lenght | change from baseline LES lenght at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in LES (Lower Esophageal Sphincter) lenght | change from baseline LES lenght at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in LES (Lower Esophageal Sphincter) IRP (Integrated Relaxation Pressure) | change from baseline LES IRP at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in LES (Lower Esophageal Sphincter) IRP (Integrated Relaxation Pressure) | change from baseline LES IRP at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in DCI (Distal Contractile Integral) | change from baseline DCI at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in DCI (Distal Contractile Integral) | change from baseline DCI at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of peristaltic waves | change from baseline rate of peristaltic waves at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of peristaltic waves | change from baseline rate of peristaltic waves at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of weak waves | change from baseline rate of weak waves at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of weak waves | change from baseline rate of weak waves at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of fragmented waves | change from baseline rate of fragmented waves at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of fragmented waves | change from baseline rate of fragmented waves at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of failed waves | change from baseline rate of failed waves at 6 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.
To identify pathophysiological factors predicting positive outcomes: changes in rate of failed waves | change from baseline rate of failed waves at 12 months
  parameter detected by High Resolution Esophageal Manometry (HRM). The manometric parameters describe the continence characteristics of the sphincter neo-valve and changes in esophageal motility after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Alberto Testoni, Professor, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- Pier Alberto Testoni, Milan, Italy

REFERENCES:
- [Derived] Testoni SGG, Cilona MB, Mazzoleni G, Fanti L, Ribichini E, Cavestro GM, Esposito D, Viale E, Notaristefano C, Zuppardo RA, Azzolini F, Passaretti S, Testoni PA. Transoral incisionless fundoplication with Medigus ultrasonic surgical endostapler (MUSE) for the treatment of gastro-esophageal reflux disease: outcomes up to 3 years. Surg Endosc. 2022 Jul;36(7):5023-5031. doi: 10.1007/s00464-021-08860-w. Epub 2021 Nov 19. PMID 34799745
- [Derived] Testoni PA, Testoni S, Mazzoleni G, Pantaleo G, Cilona MB, Distefano G, Fanti L, Antonelli M, Passaretti S. Transoral incisionless fundoplication with an ultrasonic surgical endostapler for the treatment of gastroesophageal reflux disease: 12-month outcomes. Endoscopy. 2020 Jun;52(6):469-473. doi: 10.1055/a-1124-3187. Epub 2020 Mar 18. PMID 32187630